CLINICAL TRIAL: NCT06320392
Title: CNOT7 Blood Level and Correlation to LAIR-1 in Metastatic vs Non-metastatic Breast Cancer Egyptian Patient's Cohort; a Case-Controlled Mechanistic Study
Brief Title: Implication of CCR4-NOT Complex Subunit 7 Expression in Natural Killer Cell Resistance in Metastatic Breast Cancer
Acronym: CCR4-NOT
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Prof. Nadia M. Hamdy, Ph.D., professor of biochemistry and molecular biology, Ain Shams University
Other Study IDs: RHDIRB2020110301 REC#48
Record Dates: First submitted 2024-02-23; First posted 2024-03-20 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Breast Cancer
Keywords: CNOT7; Breast cancer; Metastasis; Natural killer; LAIR-1
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — * blood samples Four milliliters of peripheral venus blood were withdrawn once from each patient, under strict sterile conditions, following standard safety procedures. Sera obtained after centrifugation were aliquoted into three clean Eppendorf tubes and stored at -80°C.
  * Parafin sections Tissue Samples The tumor was fixed in 10% neutral buffered formalin fixative for 24 hours at room temperature before being embedded in paraffin using a TissueTek VIP automated processor in accordance with the standard protocol used in the laboratory for breast tumor diagnosis and staging, Mansoura University Hospitals.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- metastatic: 44 female BC patients, volunteered in the study, diagnosed with metastatic BC. Patients were enrolled randomly from the Clinical Oncology Department, Faculty of Medicine, Mansoura University Hospitals, Mansoura University, Mansoura, Egypt, after signing the IC.
- non-metastatic: 46 female BC patients, volunteered in the study, diagnosed with primary naive (non-metastatic) invasive BC . Patients were enrolled randomly from the Clinical Oncology Department, Faculty of Medicine, Mansoura University Hospitals, Mansoura University, Mansoura, Egypt, after signing the IC.

SUMMARY:
Being a mechanistic study, this work aims to figure out "the role of the cytoplasmic mRNA deadenylase CNOT7 expressed protein on NK cell resistance in metastatic BC". In other words, to explore, whether, "CNOT7 contributes to metastasis in Egyptian female metastatic BC patient's cohort, through NK cell resistance, or not."

DETAILED DESCRIPTION:
1. Introduction 1.1. Research Problem. Breast cancer (BC) is the primary cause of cancer deaths in women (1,2). The main cause of this mortality is the metastatic spread to other organs (3). Metastasis occurs when tumor cells acquire invasive features (4) and the ability to escape from antitumor immunity; innate and adaptive immune responses important for tumor control (5,6). Major impairment of peripheral blood natural killer (NK) cell maturation and cytotoxic functions was reported to accompany BC progression (7). Several gene expression profiling studies have shown that a better outcome is associated with a strong cytotoxic infiltrate containing NK cells (8,9). These data suggest that BC progression is linked to the antitumor immune efficiency of NK cells, T-cells, and B-cells. However, how BC progression affects peripheral NK cells phenotype is not abundantly investigated.

The activity of NK cells is determined by activating and inhibitory receptors present on NK cells that are triggered during target cell (herein, tumor cell) recognition, inducing a positive or a negative cell signaling pathway, respectively. The integration of these opposite signals determines NK cell activation weight (10). Recent studies have shown that several molecules, notably inhibitory factors, often found in the tumor microenvironment (TME) can sharply impair NK cells' phenotype and functions (11,12) resulting in a decreased expression of activating NK cell receptors and an increased expression of the inhibitory receptors (like LAIR-1 that was detected previously in HCC clinical blood samples T-cytotoxic cells (13). These may promote BC progression and would correlate with the decreased immune cell cytotoxic function encountered by NK cells and T-cells or B-cells (14).

1.2. Aim and Objectives. To explore CNOT7 role related to immune cells resistance in BC metastasis, the investigators attempted to measure the serum levels of CNOT7 in Egyptian female BC patients' cohort in relation to the clinicopathological parameters. CNOT7 tissue expression in BC tissue samples categorized as metastatic vs non-metastatic tumor alongside with adjacent non-tumor tissue margin were measured. Further, quantified the inhibitory receptor on NK cells namely; LAIR-1 serum levels, whose overexpression would be linked to the aggressive BC features and adverse clinical outcome(s) (22) manifested as TNM. The correlation of CNOT7 with LAIR-1 blood levels to be assessed clinically and to be confirmed or rolled-out via bioinformatics databases search and in silico analysis. Per the investigators are looking for BC metastasis mechanism, not just exploring CNOT7 or LAIR1 blood levels, therefore, finding more therapeutic options, via CNOT7 molecular docking or through blocking its down-stream pathways or effector gene-gene networks interaction, either as potential promising treatment options. Where, these pathways and interactions will be retrieved from KEGG pathways search, further addressed through text-mined interactions or search into curated in silico bioinformatics DBs.

2.1. Study Participants 2.1.1. Ethical Approval and Informed Consent to participate. Ethical approval was obtained from Ain Shams University, Faculty of Pharmacy's review board Research Ethical Committee (REC ID# 48, October 20th, 2021).

2.1.2. The study was carried out according to guidelines by the World Medical Association (WMA) fulfilling the Declaration of Helsinki ethical principles for medical research involving human subjects, the revised July 2018 version, where all participating individuals signed the ethically approved informed consent (IC).

2.1.3. BC Patients' Groups. 90 female BC patients, volunteered in the study, diagnosed with either primary naïve (non-metastatic) invasive BC (46 patients) or metastatic BC (44 patients). Patients were enrolled randomly from the Clinical Oncology Department, Faculty of Medicine, Mansoura University Hospitals, Mansoura University, Mansoura, Egypt, after signing the IC.

2.1.4. BC diagnosis was carried out with mammogram and magnetic resonance imaging (MRI). Full history was collected and recorded for all study participants (n = 90).

Blood samples and the tissue paraffin blocks were collected for those who met the inclusion criteria and signed the IC.

2.1.5. Patients' clinical and pathological features. For all BC participants, full family disease/cancer history was recorded, as well as patients' diabetic status (yes vs no), number of pregnancies (either less or more than 2), menopausal status (pre- vs post-), and treatment(s) received (neoadjuvant chemotherapy, adjuvant chemotherapy, endocrine therapy, or mastectomy). Patients' individual current cancer status and the tumor clinical assessment, done at the Faculty of Medicine, Mansoura University Hospital, Mansoura University, using the tumor-node-metastasis (TNM) categorization according to the 8th edition of the American Joint Committee on Cancer (AJCC) staging manual and the Bloom-Richardson Scale for histological grading (24) collected from patients' data files, after a biopsy was taken at the time of BC surgical exploration/examination.

Immunohistochemistry (IHC) results for the proliferation index Ki-67 (being either low or high), estrogen receptor (ER), progesterone receptor (PR) status, and the human epidermal growth receptor 2 (HER2/neu) (each either positive or negative), body mass index (BMI) kg/m2 (normal, overweight, and obese 18.5-24.9, 25-29.9, and ≥30 kg/m2, respectively) (25), lymph node (LN) status (none N0, N1-3, N4-9, ≥ 10) (26), and age in years, were all collected from patients' files and tabulated for statistical analysis.

Molecular BC subtype (27) if luminal like (ER+ and/or PR+), HER-2 overexpression (ER-, PR-, HER-2+), or triple-negative BC (TNBC) (ER-, PR-, HER-2-) and histological BC subtypes (28) if invasive ductal carcinoma (IDC) or not, were all recorded for correlation analysis.

3. Methods 3.1. Biochemical Analysis 3.1.1. ELISA 3.1.1.1. CNOT7 ELISA CNOT7 was assessed using Human CCR4 NOT transcription complex subunit 7 (CNOT7) ELISA Kit, Mybiosource, USA, following the manufacturer's instructions. In brief, the standards and serum samples of both non-metastatic BC and metastatic BC groups were incubated together with CNOT7-HRP conjugate in an anti-CNOT7 antibody pre-coated ELISA plate supplied by the manufacturer for an hour at 37°C. After the incubation period, wells were decanted and washed five times manually using a pre-diluted wash buffer provided by the manufacturer. Wells incubated with a substrate for HRP enzyme for an hour at 37°C. Finally, a stop solution was added to stop the reaction. The color intensity produced was measured spectrophotometrically at 450 nm in a microplate reader. A standard curve was plotted relating the color intensity (Optical Density (O.D.)) to the concentration of standards. The CNOT7 concentration in each sample was interpolated from this standard curve (supplementary file).

3.1.1.2. LAIR-1 ELISA LAIR-1 was assessed using Human LAIR-1 ELISA Kit, Mybiosource, USA. Standards and samples were pipetted into the wells of an ELISA plate pre-coated with a LAIR-1 specific antibody supplied by the manufacturer. The plate was then covered and incubated at 37°C for 45 min. followed by a 5 times manual washing step using wash buffer that was previously diluted. An HRP-Conjugated detection antibody was added to the plate and it was incubated again at the same temperature for 30 min. Afterwards, the plate was washed as explained previously and incubated with chromogen solutions for 15 min. followed by a final step of adding stop solution. The intensity of color was measured spectrophotometrically at 450 nm in a microplate reader. A standard curve is plotted relating the intensity of the color (O.D.) to the concentration of standards. The LAIR-1 concentration in each sample was interpolated from this standard curve (supplementary file). Standards were prepared from a stock solution and a standard diluent provided by the manufacturer producing a 2-fold dilution series 3.1.1.3. s.Insulin ELISA Serum insulin assay was performed using Hyperion Inc., Miami, FL, USA ELISA kit. The test sample's color intensity is directly inversely related to its insulin concentration. The normal insulin adult range level is 0-25 mU/L.

3.1.2. Immunohistochemistry 3.1.2.1. CNOT7 IHC staining protocol Using paraffin sections mounted on positively charged slides using avidin-biotin- peroxidase complex (ABC) technique (29). Sections from each group were treated with CNOT7 (M01) (ABNOVA, Cat# H00029883-M01, Monoclonal antibody, Clone 2F6) at 1:25 dilution before being exposed to the chemicals necessary for the ABC method (Vectastain ABC-HRP kit, Vector laboratories). To detect antigen-antibody complexes, marker expression was tagged with peroxidase and colored with diaminobenzidine (DAB, manufactured by Sigma). Negative controls were included using non-immune serum in place of the primary or secondary antibodies. Leica microscope (CH9435 Hee56rbrugg) (Leica Microsystems, Switzerland) was used to evaluate IHC stained sections (Leica Microsystems, Switzerland).

3.1.2.2. Quantitative Evaluation of CNOT7 IHC Results "Area %" In each serial section of the analyzed patients' groups, six high power fields (x 400) with positive brown immunostaining were chosen for examination. The area% of CNOT7-stained sections was calculated using the Leica QWin 500 image analyzer computer system (UK). This image analyzer entailed a Leica microscope, a colored video camera, colored monitor and a hard disc of a Leica IBM personal computer linked to the microscope and managed by Leica QWin 500 software.

Area % data were statistically reported in terms of mean and standard error of mean (mean ± S.E.M) for eight images from four non-metastatic samples and four metastatic samples.

3.2. In silico Bioinformatics Analysis 3.2.1. Breast cancer Gene Expression Miner v5.0 (bc-GenExMiner v5.0) Updated on June 28th, 2023.

http://bcgenex.ico.unicancer.fr/BC-GEM/GEM-Accueil.php?js=1 (30) to explore the correlation between CNOT7 and LAIR1.

3.2.2. Function module of LinkedOmics used to perform analysis of Gene Ontology biological process (GO_BP) with gene set enrichment analysis (GSEA) http://www.linkedomics.org/ (31).

3.2.3. Gene-Gene interactions and pathways from in silico curated DBs and text-mining Via Genome Browser for target genes using University of California Santa Cruiz (UCSC) (32) Genomics institute http://genome.ucsc.edu/index.html LAIR1 and CNOT7 genes interactions were retrieved, with mentioning known inhibitor drug(s) from DrugBank.

3.2.4. Protein-Protein Interaction (PPI) from the Search Tool for the Retrieval of Interacting Genes/Proteins (STRING) database version 11.5 https://string-db.org/ which predicts interactions based on relevant experimental data, sequencing results, and literature from >1100 fully sequenced organism (33). Accessed on Jan. 20th, 2023, to explore LAIR-1 interacting proteins.

https://string-db.org/cgi/network?taskId=bQyD5DID27nM&sessionId=bFHqdPHoGJPF 3.2.5. Exploring Gene Expression patterns across Normal and Tumor tissues (GENT2) with survival http://gent2.appex.kr/gent2/ 3.3. Molecular Docking: 3.3.1. Preparation of the protein structures of LAIR-1 and CNOT7 https://www.protocols.io/view/protein-ligand-docking-using-moe-bnxxmfpn?step=2 From the protein data bank (PDB) https://www.rcsb.org/search the crystal structure of Human LAIR-1 (PDB ID: 3RP1) https://www.rcsb.org/structure/3RP1 After loading the structures in molecular operating environment (MOE) https://www.chemcomp.com/Products.htm Integrated Computer-Aided Molecular Design Platform, they were prepared using the default parameters in the 'QuickPrep Panel' including the removal of water molecules, adding hydrogen atoms to the protein structure, adjusting protonation states, and ensuring energy minimization of the protein structures with Amber10:EHT force field.

Since those crystal structures were not co-crystallized with any ligands, MOE SiteFinder, a program for binding-site analysis equipped in the MOE was used to predict the possible binding sites. Those pockets are ranked based on their propensity for ligand binding (PLB). CNOT7 is a receptor with no available PDB co-crystallized structure, therefore, the investigators used the MOE siteFinder tool to help in our study, with the guide of previous literatures reporting several essential amino acids residues involved in ligand-CNOT7 protein interactions like Glu247, Tyr260, Glu278 (34,35) have been identified as relatively significant.

3.3.2. Ligands dataset curation The 'builder program' implemented in MOE was used to model six ligands in the study; Vitamin E, Colchicine, Prodigiosin, Riboflavin, Telmisartan, and Pioglitazone, where all possible conformations at the physiological pH were obtained.

3.3.3. Docking simulations Docking of the obtained conformations of the six ligands was carried out using placement and refinement algorithms of MOE program. Initial docking of the molecules in the active sites used the 'Triangle Matcher' placement method and 'London dG' scoring function. Further postplacement refinement of docking poses was achieved by using 'GBVI/WSA dG' scoring method. The poses with minimum energy were used for visualization of the binding interactions as well as occupancy of the binding site of the receptors.

3.4. Statistical Analysis 3.4.1. Data collected were recorded and analyzed using the Statistical Package for Social Science software (SPSS, Version 17, Chicago, IL, USA).

3.4.2. Qualitative data were presented as frequencies (n) and percentages (%). 3.4.3. Test for quantitative data normality was performed using the Shapiro-Wilk calculator. Normally distributed variables were represented as mean ± S.E.M and analyzed using two samples independent Students' t-test for comparison of two groups. Not normally distributed data were presented as medians (interquartile ranges as first to third quartiles or 25th-75th quartiles) and analyzed using the Mann-Whitney (U) test.

3.4.4. ROC curve was performed to detect the best cut-off points to categorize CNOT7 and LAIR-1 serum levels into low and high expression subgroups.

3.4.5. The Chi-square-test was used to evaluate the association between CNOT7 serum levels and clinicopathological parameters. Pearson correlation test was used to assess the association between parametric variables. Point-biserial correlations were used to determine the correlation between parameters when one of them was a dichotomous variable.

3.4.6. The level of significance was set at P< 0.05 and confidence level (C.I) or interval at 95% and 5%, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old with breast carcinoma of no special type (NST) confirmed pathologically.

Exclusion Criteria:

* breast cancer patients with blood disorders
* breast cancer patients with any cancer other than BC
* breast cancer patients with liver cirrhosis
* breast cancer patients with uterine or urinary bladder diseases
* breast cancer patients with incomplete data or incomplete histopathology diagnosis report

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female with breast cancer (metastatic or non-metastatic)
Study Population: 90 Egyptian female BC patients, volunteered in the study, diagnosed with either primary naive (non-metastatic) invasive BC (46 patients) or metastatic BC (44 patients). Patients were enrolled randomly from the Clinical Oncology Department, Faculty of Medicine, Mansoura University Hospitals, Mansoura University, Mansoura, Egypt, after signing the IC.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Cytoplasmic mRNA deadenylase CNOT7 protein expression level in metastatic/advanced localized and non-metastatic BC sera using ELISA. | 12 months
CNOT7 tissue expression level in BC tissue samples categorized as metastatic vs non-metastatic tumor alongside with adjacent non-tumor tissue margin using immunohistochemistry. | 18 months
LAIR-1 protein expression level in BC patients peripheral blood samples using ELISA. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Hamdy, PhD, Principal Investigator — Faculty of pharmacy Ain Shams University
Locations (1):
- Faculty of Pharmacy, Ain Shams University, Advanced Biochemistry Research Lab, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided